CLINICAL TRIAL: NCT01369407
Title: REVIVE-IT Registry (REVIVAL: Registry Evaluation of Vital Information For VADs in Ambulatory Life)
Brief Title: REGISTRY EVALUATION OF VITAL INFORMATION FOR VADs IN AMBULATORY LIFE
Acronym: REVIVAL
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Keith Aaronson, Bertram Pitt M.D. Collegiate Professor of Cardiovascular Medicine and Professor of Internal Medicine, Medical School, University of Michigan
Other Study IDs: REVIVE-IT REGISTRY (REVIVAL); HHSN268201100026C (Other Grant/Funding Number: NHLBI)
Record Dates: First submitted 2011-06-01; First posted 2011-06-08 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Congestive Heart Failure
Keywords: Heart failure; HF; Heart Diseases; Cardiovascular Diseases; Heart Failure NYHA class III; Advanced heart failure; Systolic Heart Failure
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases; Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Biomarker Samples will be collected at the Baseline B assessment. Samples for Genomic Analysis will be collected at the Baseline B visit for subjects that consented to collection of this sample type.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Enrolled Subjects: Enrolled subjects participate for up to 2 years
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Not an interventional study

SUMMARY:
REVIVAL will establish a prospective, observational, multicenter patient cohort in ambulatory patients with chronic, advanced, systolic heart failure that will provide a greater understanding of their clinical trajectory (rates of hospitalizations, transplantation, MCSD use and death), and of how baseline clinical risk measures are related to prognosis.

DETAILED DESCRIPTION:
REVIVAL will establish a prospective, observational, multicenter patient cohort in ambulatory patients with chronic, advanced, systolic heart failure that will provide a greater understanding of their clinical trajectory (rates of hospitalizations, transplantation, MCSD use and death), and of how baseline clinical risk measures are related to prognosis. Within the broader goal of 1) improving prognostic assessment in chronic, ambulatory, advanced systolic heart failure, additional targeted goals are to 2) better inform the selection of appropriate candidates for a future study of a strategy of early LVAD therapy vs. optimal medical management in this population, and 3) determine the feasibility of identifying candidates for such a trial. Therefore, the target population will have known high-risk features for increased mortality and hospitalization (e.g., frequent hospitalization, reduced exercise capacity, elevated BNP or N-terminal proBNP, increased Seattle Heart Failure Model risk score, reduced Heart Failure Survival Score).

The REVIVE-IT Registry (i.e., REVIVAL) is a prospective cohort study to be conducted in up to twenty five (25) participating Clinical Sites in the USA. The study will continue until up to 400 eligible heart failure heart failure subjects have been enrolled (estimated length of accrual is 12 months).

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory.
2. Chronic systolic heart failure ≥ 12 months.
3. NYHA II - IV for at least 45 of the last 60 days.
4. Last documented left ventricular ejection fraction ≤ 35% by any imaging modality.
5. Age 18 - 80 years.
6. Under the care of a cardiologist at study site.
7. On appropriate evidenced -based heart failure medications - ACE inhibitor, ARB or sacubitril/valsartan [LCZ-696]; beta blocker; aldosterone antagonist; hydralazine/long-acting nitrate [required of African-American subjects only] for ≥ 3 months absent contraindications or intolerances.
8. Has ICD or CRT-D. If CRT-D, present for ≥ 3 months.
9. Demonstrated advanced heart failure, including any one of the following*:

   i. Serum sodium ≤ 135 mEq/L (obtained as an outpatient)** ii. Serum BNP ≥ 750 pg/mL or NT-proBNP ≥ 3000 pg/mL** (obtained as an outpatient) iii. Seattle Heart Failure Model (SHFM) one year predicted survival ≤ 85%** iv. Heart Failure Survival Score (HFSS) ≤ 7.19** v. Peak VO2 ≤ 55% of predicted for age by Wasserman equation or ≤ 14 ml/kg/min, with RER ≥ 1.05*** vi. VE/VC02 slope > 40*** vii. 6 minute walk test (6MWT) distance ≤ 350 m without significant non-cardiac limitation** viii. Currently listed as Heart Transplant Status II due to heart failure limitation

   Or

   History of one (1) hospitalization (≥ 24 hours) for acute or acute on chronic heart failure in the past year with additional history to include:

   i. Serum BNP ≥ 500 pg/mL or NT-proBNP ≥ 2000 pg/mL** (obtained as an outpatient)

   Or

   History of two (2) hospitalizations (≥ 24 hours) for acute or acute on chronic heart failure in the past year.

   * Qualifying measure must be the most recent of that type of measure obtained (i.e., a BNP ≥ 1000 obtained 2 months prior would not qualify the heart failure subject if a more recent BNP was < 1000)

   **Using values obtained within the prior 90 days, except for peak VO2 within 365 days

   ***Obtained within the prior 365 days
10. Willingness to continue to receive heart failure care from the enrolling advanced heart failure clinic over the next two (2) years and to come for all scheduled study visits.

12. Written Informed consent given.

Exclusion Criteria:

1. Known serious medical problem other than heart failure that would be expected to limit 2-year survival (≥50% mortality within 2 years from non-heart failure diagnosis).
2. Patient is not likely to be compliant with the protocol, in the opinion of the Investigator.
3. Currently hospitalized.
4. Current use of an intravenous inotrope.
5. Primary functional limitation from non-cardiac diagnosis even if not likely to limit survival.
6. Chronic hemodialysis or peritoneal dialysis or a serum creatinine value of ≥ 3 mg/dL at time of enrollment.
7. Cardiac amyloidosis, cardiac sarcoidosis, constrictive pericardial disease, active myocarditis or congenital heart disease with significant structural abnormality.
8. Hypertrophic cardiomyopathy unless dilated LV and no outflow gradient.
9. Cardiac conditions that are amenable to surgical or percutaneous procedures (other than VAD or transplant) that would substantially improve prognosis and for which this subject is a reasonable candidate, regardless of whether the procedure will or will not be performed.
10. Uncorrected hyperthyroidism or hypothyroidism.
11. Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical records should be reviewed to assess for potential enrollment into the REVIVE-IT Registry. Heart failure subjects that meet all criteria should be approached to consent for this study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
To characterize clinical outcomes, quality of life and functional impairment over two (2) years in a population of ambulatory patients on evidence-based therapy with advanced chronic systolic heart failure who may benefit from VAD therapy | 2 years
To evaluate the relationship between heart failure subject's modeled prognosis, self assessed prognosis, preferences for end of life care and thresholds for considering VAD implant. | 2 years
To evaluate caregiver burden associated with heart failure subject's measures of heart failure severity, quality of life, functional limitations and with preferences for care and thresholds for considering device implant. | 2 years.
To determine health-associated costs for heart failure subjects in the registry. | 2 years.
To provide the REVIVE-IT Registry to the INTERMACS study group to be used in comparative analyses of outcomes of patients treated with medical versus VAD therapy. | 2 years.

SECONDARY OUTCOMES:
Hospitalization | 2 years
  Assessed throughout participation
Stroke | 2 years
  Assessed throughout participation
MCSD | 2 years
  Assessed throughout participation (study endpoint)
Transplant | 2 years
  Assessed throughout participation (study endpoint)
Death | 2 years
  Assessed throughout participation

CONTACTS AND LOCATIONS:
Overall Officials: Keith Aaronson, MD, MS, Principal Investigator — University of Michigan; Garrick Stewart, MD, Principal Investigator — Brigham and Women's Hospital; Doug Mann, MD, Study Chair — University of Washington - St. Louis
Locations (21):
- United States (21):
  - University of Alabama, Birmingham, Alabama
  - Cedars-Sinai Medical Care Foundation, Beverly Hills, California
  - University of Colorado, Denver, Aurora, Colorado
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University, St. Louis, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - INTEGRIS, Oklahoma City, Oklahoma
  - Abington Jefferson Health, Abington, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UT Southwestern, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Inova Heart and Vascular Institute, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Aaronson KD, Stewart GC, Stevenson LW, Richards B, Khalatbari S, Cascino TC, Ambardekar AV, Stehlik J, Lala A, Kittleson MM, Palardy M, Mountis MM, Pagani FD, Jeffries N, Taddei-Peters WC, Mann DL; REVIVAL Investigators. Optimizing Triage of Ambulatory Patients With Advanced Heart Failure: 2-Year Outcomes From REVIVAL. JACC Heart Fail. 2024 Oct;12(10):1734-1746. doi: 10.1016/j.jchf.2024.05.008. Epub 2024 Jul 3. PMID 38970587
- [Derived] Cascino TM, Colvin MM, Lanfear DE, Richards B, Khalatbari S, Mann DL, Taddei-Peters WC, Jeffries N, Watkins DC, Stewart GC, Aaronson KD; REVIVAL Investigators. Racial Inequities in Access to Ventricular Assist Device and Transplant Persist After Consideration for Preferences for Care: A Report From the REVIVAL Study. Circ Heart Fail. 2023 Jan;16(1):e009745. doi: 10.1161/CIRCHEARTFAILURE.122.009745. Epub 2022 Oct 19. PMID 36259388
- [Derived] Lala A, Shah KB, Lanfear DE, Thibodeau JT, Palardy M, Ambardekar AV, McNamara DM, Taddei-Peters WC, Baldwin JT, Jeffries N, Khalatbari S, Spino C, Richards B, Mann DL, Stewart GC, Aaronson KD, Mancini DM; REVIVAL Investigators. Predictive Value of Cardiopulmonary Exercise Testing Parameters in Ambulatory Advanced Heart Failure. JACC Heart Fail. 2021 Mar;9(3):226-236. doi: 10.1016/j.jchf.2020.11.008. Epub 2021 Feb 3. PMID 33549559
- [Derived] Cascino TM, Kittleson MM, Lala A, Stehlik J, Palardy M, Pamboukian SV, Ewald GA, Mountis MM, Horstmanshof DA, Robinson SW, Shah P, Jorde UP, McLean RC, Richards B, Khalatbari S, Spino C, Taddei-Peters WC, Grady KL, Mann DL, Stevenson LW, Stewart GC, Aaronson KD; REVIVAL Investigators. Comorbid Conditions and Health-Related Quality of Life in Ambulatory Heart Failure Patients: REVIVAL (Registry Evaluation of Vital Information for VADs in Ambulatory Life REVIVAL). Circ Heart Fail. 2020 May;13(5):e006858. doi: 10.1161/CIRCHEARTFAILURE.119.006858. Epub 2020 May 18. PMID 32418478
- [Derived] Pagani FD, Aaronson KD, Kormos R, Mann DL, Spino C, Jeffries N, Taddei-Peters WC, Mancini DM, McNamara DM, Grady KL, Gorcsan J 3rd, Petrucci R, Anderson AS, Glick HA, Acker MA, Eduardo Rame J, Goldstein DJ, Pamboukian SV, Miller MA, Timothy Baldwin J; REVIVE-IT Investigators. The NHLBI REVIVE-IT study: Understanding its discontinuation in the context of current left ventricular assist device therapy. J Heart Lung Transplant. 2016 Nov;35(11):1277-1283. doi: 10.1016/j.healun.2016.09.002. Epub 2016 Oct 6. PMID 27836022